CLINICAL TRIAL: NCT04612569
Title: Feasibility and Impact of a Trimodal Prehabilitation and Rehabilitation Program to Reduce the Predicted Low Anterior Resection Syndrome After Radical Rectal Cancer Treatment. A Non-Randomized Prospective Study Phase II. PRELARS Study
Brief Title: Feasibility and Impact of a Prehabilitation and Rehabilitation Program for the Continuity of Care in Severe Low Anterior Resection Syndrome.
Acronym: PRELARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Donostia (Other)
Responsible Party: Principal Investigator, Prof. Jose M Enríquez-Navascués, PhD; Head of service, Hospital Donostia
Other Study IDs: ELO-PRE-2020-01
Record Dates: First submitted 2020-10-12; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Rectal Cancer; Low Anterior Resection Syndrome; Faecal Incontinence
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome; Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with sphincter saving procedures of rectal cancer usually experience intestinal dysfunction, including difficulty emptying the bowel and faecal incontinence, leading to a detriment in the quality of life. A prospective study is proposed to measure de feasibility and the impact of a continuous care programme for the prevention or reduction of intestinal dysfunction disorders. The intervention lies on prehabilitation and rehabilitation with physiotherapy, biofeedback and neuromodulation, is assisted by a telematic information system (APP for the monitoring of education on physiotherapy and surveillance).

DETAILED DESCRIPTION:
-Study design: A single-arm, non-randomized prospective study that will initially evaluate the compliance and feasibility of a prehabilitation and / or functional rehabilitation program in patients with anterior rectal resection with mesorectal excision for rectal cancer. In addition, clinical outcome variables will be obtained to evaluate the possibility of a subsequent efficacy study.

-Patient selection: Participation in this study will be proposed to all consecutive patients with rectal cancer who are expected to perform a low anterior resection of the rectum with mesorectal excision and colorectal anastomosis with or without protective ileostomy, older than 18 years, who give their informed consent, and who can carry out a pelvic floor physiotherapy program and be susceptible to tibial neurostimulation.

Exclusion criteria will be a POLARS score less than 20 (LARS-minor or non-LARS), the existence of residual or distant locoregional disease, the presence of inflammatory bowel disease (IBD), a previous known diagnosis of irritable bowel syndrome (IBS) , patients with intestinal resections other than the rectum, existence of anastomotic complications, or inability to perform pelvic muscle physiotherapy, presence of trophic disorders in the ankles (post-febile syndrome), known diabetic neuropathy, carriers of pacemakers or implantable defibrillators, and with previous SNS or PTNS.

-Interventions:

The package of interventions consists on:

1. Educational session: colorectal nursing consultation, in which the inclusion / exclusion criteria are checked, the preoperative data relative to the outcome measures scales (POLARS, Vaizey and QLQ-C30) and the pre and postoperative clinical variables are filled in of interest to the study.

   After explaining the components, phases and duration of the prehabilitation or rehabilitation program, the informed consent of the patients is obtained.

   In this first visit, the pelvic floor muscle rehabilitation exercises to be performed are shown and supervised, recording the baseline data of the modified Oxford scale and the PERF scheme (Power, Endurance, Repetition, Fast).
2. Pelvic Floor Physical Therapy (FTSP) and Biofeedback: Patients will complete three sets of muscle exercises per day: slow pelvic floor contractions, maximum sustained contractions, and rapid pelvic floor contractions; performing 10 repetitions of each modality per series, with an approximate duration of 2-3 minutes each. These exercises can be performed in any position, moment or circumstance at the convenience of the patients.

   At each visit to the nursing consultation, the exercises will be supervised and on specific dates (see program diagram) the contraction force will be quantified using the modified Oxford scale, the PERF scheme and an anal manometry.

   For anal manometry, the Anopress device (THD SpA, Correggio (RE), Italy) will be used, a portable and wireless manometer that uses high resolution air to fill the probes that register pressures generated in the anal canal. A standard protocol was followed for all patients. Resting pressure data are recorded, with voluntary contractions, involuntary contractions (eg, with coughing) and resistance pressures (the duration of up to 50% of the maximum effort pressure is defined in a maximum of ten seconds). A second catheter with a distensible balloon is used to measure rectal sensitivity to distension and the inhibitory anorectal reflex. There will be 2 biofeedback sessions.

   As controls of adherence to the program, patients will keep either a diary with the exercises performed or the records of the pelvic floor exercise program app.
3. Percutaneous neurostimulation of the posterior tibial nerve: For the PTNS, an Urgent PC® device (Uroplasty, NL) is used; the procedure will be performed in outpatient consultations by colorectal nurses, following the standard technique recommended by the manufacturer. Stimulation is carried out using a 34 G needle electrode inserted at a cranial point 3-4 cm and 2 cm posterior to the medial malleolus, and another adhesive electrode near the arch of the foot of the same leg. The electrostimulation parameters are as follows: a pulse width of 200 ms, a frequency of 20 Hz, and an increased current until flexion of the fingers was first noticed (0-18 mA). The program includes a total of 20 sessions of 30 minutes each, once a week for 12 consecutive weeks, followed by 4 additional sessions once every 15 days for the next 2 months and 4 additional sessions once a month.
4. APP that allows physiotherapy education and monitoring of results.

   * Clinical variables and outcome measures:

The outcome measures will be the POLARS predictive score of the LARS, Vaizey (St. Mark's) of fecal incontinence and the EORTC QLQ-30 of quality of life, obtained perioperatively, and the LARS, Vayzey and QLQ-30 scales at 6 months and year of surgery or closure of the protective stoma. As measurements of the FTSP, the results of the anal manometries, the modified Oxford scale and the PERF scheme will be obtained. Adherence to the FTSP program will be evaluated by the percentage of compliance with the exercises according to the patients' diary or from the records of the pelvic floor app.

To assess the degree of acceptability to the program, the percentage of patients who leave it voluntarily, totally or partially, will be evaluated, as well as using a visual analog scale (VAS) obtained at the end of the program.

The following data will be recorded as clinical variables: 1) sex; 2) age; 3) BMI; 4) date of rectal resection; 5) performance or not of protection stoma and, where appropriate, date of stoma closure; 6) administration or not of radiochemotherapy or neoadjuvant short-course radiotherapy; 7) Height of tumor measured by MRI; 8) Open, laparoscopic, taTME or mixed approach (abdominal part by laparoscopy and open pelvic part); 9) Total or partial mesorectal excision; 10) Quality of mesorectal resection; 11) Height of the anastomosis (from anal margin); 12) type of anastomosis (manual or mechanical, end-to-end or lateral-end or pouch-end); 13) Administration of adjuvant chemotherapy; 14) Postoperative complications according to the Clavien-Dindo classification; 15) Postoperative staging; and 16) Astringent medication, forming fecal mass or hygienic-dietary modifications throughout the study.

RESULTS:

The feasibility and adherence to the program will be initially analyzed through the percentage of compliance with the PTNS sessions and the proposed FSTP exercises performed in the first 15 cases, in order to be able to adjust the program scheme and estimate a representative sample size.

The main objective of the study will be to compare the estimated preoperative LARS score (POLARS) with the postoperative LARS score observed at 6 months and one year after radical surgery (or closure of the ileostomy) for rectal cancer, considering it as clinically relevant descending at least one category from POLARS- major to LARS- minor (or not LARS) in at least 50% of patients. Secondary objectives will be to assess the effect of the interventions on fecal incontinence (Vaizey), quality of life (QLQ-C30) and pelvic floor contractility (anal manometry, Oxford scale and PERF).

ELIGIBILITY:
Inclusion Criteria:

* Low anterior resection of the rectum with mesorectal excision and colorectal anastomosis with or without protective ileostomy
* POLARS score >20
* over 18 years of age
* give their informed consent
* Patients who can perform a pelvic floor physiotherapy program and to tibial nerve stimulation.

Exclusion Criteria:

* POLARS score less than 20
* LARS-minor or non-LARS
* The existence of residual or distant locoregional disease
* Inflammatory bowel disease (IBD)
* A previous known diagnosis of irritable bowel syndrome (IBS)
* Intestinal resections other than the rectum
* Existence of anastomotic complications
* Inability to perform pelvic muscle physiotherapy, presence of trophic disorders in the ankles (post-febile syndrome)
* Known diabetic neuropathy
* Carriers of pacemakers or implantable defibrillators, and patients who are have previously performed SNS or PTNS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer who are expected to undergo a low anterior resection of the rectum with mesorectal excision and colorectal anastomosis with or without protective ileostomy, older than 18 years, who give their informed consent, and who can carry out a pelvic floor physiotherapy program and be susceptible to tibial neurostimulation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Impact of a multimodal package of prehabilitation and rehabilitation in patients with low anterior resection syndrome | October 2020- September 2021
  To analyze the feasibility of the introduction of a multimodal package of integrated interventions (educational, pelvic floor physiotherapy, biofeedback and posterior tibial neurostimulation-PTNS-) with the objective of reducing the severity of predictable intestinal dysfunction after the radical surgery for rectal cancer, measured by the number of patients that complete the treatment.

SECONDARY OUTCOMES:
Feasibility of introduction of APP for the education and follow-up | October 2020- September 2021
  Compliance comprehensive outpatient therapeutic program, supported by the introduction of an APP device; measured by the proportion of patients that use the APP and the use that gives each patient.
Assessment of the improvement of scores in faecal incontinence, | October 2020- September 2021
  To assess the effect of multimodal interventions on aspects of fecal incontinence, measured by the Vaizey Faecal Incontinence score (Vaizey Score 0-24; 0 perfect continence and 24 is total incontinence).
Analysis of the correlation between estimated POLARS score and postoperative LARS score | October 2020- September 2021
  To analyze the correlation between the estimated preoperative POLARS score and the postoperative LARS score collected at 6 months and one year after radical surgery or closure of the derivative stoma. (LARS score 0-42; 0-20 No LARS; 21-29 Minor LARS; 30-42 Major LARS)
Assessment of the improvement of quality of life | October 2020- September 2021
  To assess the effect of multimodal interventions on aspects of quality of life, measured by the EORTC QLQ-30 quality of life score (0-100; higher measures mean better quality of life).
Assessment of the improvement of pelvic floor contractility | October 2020- September 2021
  To assess the effect of multimodal interventions on pelvic floor contractility with the results of anal manometries, the modified Oxford scale (0-5; 0 means No contraction and 5 means Strong contraction).

CONTACTS AND LOCATIONS:
Locations (1):
- Garazi Elorza, San Sebastián, Guipuzcoa, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012 May;255(5):922-8. doi: 10.1097/SLA.0b013e31824f1c21. PMID 22504191
- [Background] Enriquez-Navascues JM, Labaka-Arteaga I, Aguirre-Allende I, Artola-Etxeberria M, Saralegui-Ansorena Y, Elorza-Echaniz G, Borda-Arrizabalaga N, Placer-Galan C. A randomized trial comparing transanal irrigation and percutaneous tibial nerve stimulation in the management of low anterior resection syndrome. Colorectal Dis. 2020 Mar;22(3):303-309. doi: 10.1111/codi.14870. Epub 2019 Oct 21. PMID 31585495
- [Background] Battersby NJ, Bouliotis G, Emmertsen KJ, Juul T, Glynne-Jones R, Branagan G, Christensen P, Laurberg S, Moran BJ; UK and Danish LARS Study Groups. Development and external validation of a nomogram and online tool to predict bowel dysfunction following restorative rectal cancer resection: the POLARS score. Gut. 2018 Apr;67(4):688-696. doi: 10.1136/gutjnl-2016-312695. Epub 2017 Jan 23. PMID 28115491
- [Background] Altomare DF, Picciariello A, Ferrara C, Digennaro R, Ribas Y, De Fazio M. Short-term outcome of percutaneous tibial nerve stimulation for low anterior resection syndrome: results of a pilot study. Colorectal Dis. 2017 Sep;19(9):851-856. doi: 10.1111/codi.13669. PMID 28371160
- [Background] Lee KH, Kim JS, Kim JY. Efficacy of biofeedback therapy for objective improvement of pelvic function in low anterior resection syndrome. Ann Surg Treat Res. 2019 Oct;97(4):194-201. doi: 10.4174/astr.2019.97.4.194. Epub 2019 Oct 1. PMID 31620393